CLINICAL TRIAL: NCT01377506
Title: Translation of Obesity and Cognitive Research in a Rural State Via Senior Centers
Brief Title: Translation of Obesity and Cognitive Program by Lay Health Educators
Acronym: Coaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104877; R18DP001145 (NIH)
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Overweight; Memory Disorder
Keywords: behavioral weight control; lifestyle intervention; memory training; cognitive training; community-based
MeSH Terms: conditions — Overweight; Memory Disorders | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Diabetes Prevention Program Lifestyle Balance Intervention delivered by lay health educator
  Interventions: Behavioral: lifestyle counseling
- Cognitive Training (Active Comparator): Adaptation of SeniorWise Memory Training program for delivery by lay health educator, matched in duration and contact to the other study arm
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: lifestyle counseling — 21 session group-based behavioral weight management program delivered in senior center over 12 months by lay health educators
  Other Names: DPP Lifestyle Balance Program
  Arms: Lifestyle counseling
Behavioral: Cognitive Training — 21 session group-based cognitive training program delivered in senior center over 12 months by lay health educators
  Arms: Cognitive Training

SUMMARY:
Obesity is a major public health problem among older adults, with 31% of non-institutionalized older persons (60 years+) in the US obese and projections indicating that this will rise to 40% by 2010. A second public health challenge on the horizon for the aging US population is the increasing number of individuals experiencing cognitive decline, dementia or Alzheimer 's disease. Recent clinical trials have demonstrated efficacy in reducing risks associated with both of these significant and increasingly pervasive health problems, which are more common among rural, low income and ethnic minority populations. The Diabetes Prevention Program (DPP) Lifestyle Intervention produced sustained weight losses in a large, diverse population of high-risk individuals and dramatically reduced rates of type 2 diabetes onset, particularly among older adults. SeniorWISE produced improvements in memory in community dwelling older persons. Transferring these exciting technologies to community settings where they can benefit older adults is a pressing public health need. Therefore, the current project seeks to transfer these two evidence-based interventions to older adults in a rural state using senior centers as the venue for dissemination and lay health educators to deliver the interventions. Senior centers are a particularly attractive context for translation of evidence-based health promotion technologies in predominantly rural states like Arkansas because they have a well-established infrastructure in communities and share a common goal of promoting healthy aging and reducing health care costs. The 3-year randomized, controlled trial will evaluate translation of the interventions by randomizing senior centers (N=16) across Arkansas to implement either (1) the DPP Lifestyle Weight Loss Program or (2) the SeniorWISE Cognitive Training Program. Older (age > 60) adults (N=288) nested within senior centers will receive the programs delivered in a group format by a trained lay health educator. Primary outcomes are changes in body weight and cognitive functioning at 12 months. The multi-level evaluation plan will characterize reach, effectiveness, adoption, implementation and maintenance of the interventions, with a cost effectiveness component.

ELIGIBILITY:
Inclusion Criteria for senior centers (unit of randomization):

* located in the state of Arkansas
* agree to be randomized
* able to identify two or three volunteers or staff members willing to be trained (including IRB certification) and deliver the programs within the senior center over the course of a year
* have adequate space for group meetings and for private data collection visits
* agreement that it would be likely that they could identify 18 interested and eligible (obese and not cognitively impaired) senior adults willing to attend the program over the course of 12 months

Exclusion Criteria:

* inability to identify and secure lay health educator from within their community
* concerns of inability to recruit the requisite 18 senior adult participants who met minimal inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
weight loss | 4 and 12 month
  weight change from baseline in kg and percent weight loss [1-(12-month weight/baseline weight)

SECONDARY OUTCOMES:
cognitive function | 4 and 12 month
  change in memory (immediate and delayed) and attention

CONTACTS AND LOCATIONS:
Overall Officials: Delia S West, PhD, Principal Investigator — University of Arkansas

REFERENCES:
- [Derived] West DS, Bursac Z, Cornell CE, Felix HC, Fausett JK, Krukowski RA, Lensing S, Love SJ, Prewitt TE, Beck C. Lay health educators translate a weight-loss intervention in senior centers: a randomized controlled trial. Am J Prev Med. 2011 Oct;41(4):385-91. doi: 10.1016/j.amepre.2011.06.041. PMID 21961465